CLINICAL TRIAL: NCT06019598
Title: Licorice and Home Blood Pressure, Additional Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Peder af Geijerstam, Principal investigator, Linkoeping University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: licorice2023_additional
Record Dates: First submitted 2023-08-25; First posted 2023-08-31 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Hypertension,Essential
MeSH Terms: conditions — Essential Hypertension | interventions — Glycyrrhiza glabra extract

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Licorice (Experimental): 2 weeks of licorice corresponding to 20 mg of glycyrrhizic acid followed by 2 weeks of licorice corresponding to 50 mg of glycyrrhizic acid.
  Interventions: Other: Licorice

INTERVENTIONS:
Other: Licorice — Ecologic sweet licorice pastilles made from Glycyrrhiza glabra grown in Calabria, Italy, with a GA content of 29.9 ±2.0 mg/g.

SUMMARY:
Out-of-office blood pressure is more strongly associated with cardiovascular risk than office blood pressure. Licorice is known to raise blood pressure, but no previous studies have measured the effects on home blood pressure. The aim of this study is to analyze the association between licorice intake and home blood pressure.

DETAILED DESCRIPTION:
For a detailed background, please see Clinical Trials registration number NCT05661721. In brief, out-of-office blood pressure is more strongly associated with cardiovascular risk than office blood pressure. Licorice is known to raise blood pressure, but no previous studies have measured the effects on home blood pressure. In a previous study, the response to licorice intake varied between participants. The aim of this study is to analyze the response of the most "licorice sensitive" quartile of participants from the original study to lower dosages of licorice, corresponding to 20 and 50 milligram och GA daily.

ELIGIBILITY:
Inclusion Criteria:

* Previous participation in the Licorice and home blood pressure study (NCT05661721).

Exclusion Criteria:

* Known hypertension, cardiovascular disease, kidney disease, liver disease, hormonal disease, peanut allergy, eating disorder or headache disease (including tension headache and migraine)
* Known alcohol abuse or drug abuse (including cannabis and anabolic steroids) treatment with hormonal drugs (including oral contraceptives
* Known intolerance to licorice intake.

Ages: 18 Years to 31 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2023-09-19 (Actual); Primary Completion 2024-02-24 (Actual); Study Completion 2024-08-13 (Actual)

PRIMARY OUTCOMES:
Systolic home blood pressure | 3 days before interventions and 28 days during intervention
  Systolic home blood pressure

SECONDARY OUTCOMES:
Diastolic home blood pressure | 3 days before interventions and 28 days during intervention
  Diastolic home blood pressure
Body weight | Day 0, 14 and 28
  Body weight
Plasma sodium | Day 0, 14 and 28
  Plasma sodium
Plasma potassium | Day 0, 14 and 28
  Plasma potassium
Plasma creatinine | Day 0, 14 and 28
  Plasma creatinine
Plasma N-terminal pro B-type natriuretic peptide | Day 0, 14 and 28
  Plasma N-terminal pro B-type natriuretic peptide
Plasma renin | Day 0, 14 and 28
  Plasma renin
Serum aldosterone | Day 0, 14 and 28
  Serum aldosterone

CONTACTS AND LOCATIONS:
Overall Officials: Fredrik H Nyström, MD, PhD, Study Director — Linkoeping University
Locations (1):
- Cityhälsan Centrum, Norrköping, Östergötland County, Sweden

IPD SHARING:
Plan to Share IPD: Yes
As specified below.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: After publication in a peer-reviewed journal and for the period of time for which local archive regulations stipulate.
Access Criteria: To be determined on a case by case basis.

REFERENCES:
- [Background] Williams B, Mancia G, Spiering W, Agabiti Rosei E, Azizi M, Burnier M, Clement DL, Coca A, de Simone G, Dominiczak A, Kahan T, Mahfoud F, Redon J, Ruilope L, Zanchetti A, Kerins M, Kjeldsen SE, Kreutz R, Laurent S, Lip GYH, McManus R, Narkiewicz K, Ruschitzka F, Schmieder RE, Shlyakhto E, Tsioufis C, Aboyans V, Desormais I; Authors/Task Force Members:. 2018 ESC/ESH Guidelines for the management of arterial hypertension: The Task Force for the management of arterial hypertension of the European Society of Cardiology and the European Society of Hypertension: The Task Force for the management of arterial hypertension of the European Society of Cardiology and the European Society of Hypertension. J Hypertens. 2018 Oct;36(10):1953-2041. doi: 10.1097/HJH.0000000000001940. PMID 30234752
- [Background] Deutch MR, Grimm D, Wehland M, Infanger M, Kruger M. Bioactive Candy: Effects of Licorice on the Cardiovascular System. Foods. 2019 Oct 14;8(10):495. doi: 10.3390/foods8100495. PMID 31615045
- [Background] Parati G, Stergiou GS, Bilo G, Kollias A, Pengo M, Ochoa JE, Agarwal R, Asayama K, Asmar R, Burnier M, De La Sierra A, Giannattasio C, Gosse P, Head G, Hoshide S, Imai Y, Kario K, Li Y, Manios E, Mant J, McManus RJ, Mengden T, Mihailidou AS, Muntner P, Myers M, Niiranen T, Ntineri A, O'Brien E, Octavio JA, Ohkubo T, Omboni S, Padfield P, Palatini P, Pellegrini D, Postel-Vinay N, Ramirez AJ, Sharman JE, Shennan A, Silva E, Topouchian J, Torlasco C, Wang JG, Weber MA, Whelton PK, White WB, Mancia G; Working Group on Blood Pressure Monitoring and Cardiovascular Variability of the European Society of Hypertension. Home blood pressure monitoring: methodology, clinical relevance and practical application: a 2021 position paper by the Working Group on Blood Pressure Monitoring and Cardiovascular Variability of the European Society of Hypertension. J Hypertens. 2021 Sep 1;39(9):1742-1767. doi: 10.1097/HJH.0000000000002922. PMID 34269334
- [Background] Spinks EA, Fenwick GR. The determination of glycyrrhizin in selected UK liquorice products. Food Addit Contam. 1990 Nov-Dec;7(6):769-78. doi: 10.1080/02652039009373939. PMID 2079112
- [Background] Rizzato G, Scalabrin E, Radaelli M, Capodaglio G, Piccolo O. A new exploration of licorice metabolome. Food Chem. 2017 Apr 15;221:959-968. doi: 10.1016/j.foodchem.2016.11.068. Epub 2016 Nov 17. PMID 27979300